CLINICAL TRIAL: NCT03456375
Title: Correlation Between Serum Progesterone Levels and the Endometrial Gene Expression Profile of 238 Genes Related With Endometrial Receptivity (Through Patented ERA Test), as Well as Correlation With Endometrial Progesterone Levels.
Brief Title: Serum and Uterine Progesterone Levels and ERA Test.
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 1706-VLC-051-EL
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Endometrial Receptivity
Keywords: progesterone; artificial endometrial preparation cycle; endometrial receptivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endometrial biopsies, Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since the implantation is related with endometrial receptivity, the patient specific plasma progesterone concentration influences this pattern.

Following this hypothesis, the study establishes a correlation between the serum progesterone measured on the day of the endometrial biopsy and the endometrial receptivity with the ERA test.

DETAILED DESCRIPTION:
In patients who have had problems of assisted reproduction it is essential to establish the factors that contribute to the success of a cycle: correcting these factors means increasing the possibility of the cycle culminating in pregnancy.

In patients with embryonic implantation failures, a prevalence of non-receptive endometrium has been described after performing the ERA test of around 20%. On the other hand, a study that shows embryonic generation values below a certain threshold (25th percentile), presents a rate of evolutionary clinical gestation and lower embryo implantation.

It is logical to think that progesterone levels are lower than the state of endometrial receptivity, since the hormone is responsible for the endothelial changes that prepare the uterus for implantation. It is ERA. The result of this study is the result of the evaluation of the lifetime of the endometrial biopsy is related to the result of the same.

If desired, the determination of the probability of the day of the transfer is predictive of the pregnancy rate through the impact that the hormone has on the endometrial receptivity. This would allow to decide in the same cycle, if the patient should be in a transfer to another dimension, or should it defer to another cycle where obtain the optimal values of progesterone.

Nowadays, there are no publications in the literature that have related the concentration of progesterone with endometrial receptivity through ERA. This is the first prospective study that analyzes this relationship.

The ERA test has been chosen for the evaluation of endometrial receptivity, which is a tool that has been widely used and used in the usual clinical practice of our clinic.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women <50 years
* One or more failed IVF treatments
* Undergoing an artificial endometrial preparation cycle with hormonal replacement therapy in order to perform an endometrial receptivity analysis through ERA test.
* Endometrial thickness after estrogen treatment > 6.5 mm with trilaminar structure

Exclusion Criteria:

* Uterine alterations (fibroids, polyps or Müllerian abnormalities)
* Adnexal pathology

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile patients with background of failed IVF cycles in which an endometrial receptivity test (ERA test) is performed in the context of an artificial cycle.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Progesterone plasma levels and Endometrial receptivity analysis result | 7 months
  To evaluate correlation between progesterone plasma levels and endometrial receptivity through ERA test in infertile women.

SECONDARY OUTCOMES:
Relationship between progesterone levels in uterus and in plasma | 8 months
  To evaluate correlation between progesterone uterine levels and progesterone plasma levels

OTHER OUTCOMES:
Relationship between progesterone uterine levels and Endometrial receptivity | 8 months
  To evaluate correlation between progesterone uterine levels and endometrial receptivity through ERA test.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Labarta, MD, Principal Investigator — IVI Vakencia
Locations (1):
- IVI RMA Valencia, Valencia, Spain

REFERENCES:
- [Derived] Labarta E, Sebastian-Leon P, Devesa-Peiro A, Celada P, Vidal C, Giles J, Rodriguez-Varela C, Bosch E, Diaz-Gimeno P. Analysis of serum and endometrial progesterone in determining endometrial receptivity. Hum Reprod. 2021 Oct 18;36(11):2861-2870. doi: 10.1093/humrep/deab184. PMID 34382075